CLINICAL TRIAL: NCT06956144
Title: Exploring the Clinical Application Value of CAIX-Targeted PET Imaging in Renal Cancer Patients
Status: Recruiting | Type: Observational
Sponsor: The First Affiliated Hospital of Xiamen University (Other)
Responsible Party: Sponsor
Other Study IDs: XMFHIIT-2025SL048
Record Dates: First submitted 2025-04-25; First posted 2025-05-02 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-04

CONDITIONS: Tumor; Carbonic Anhydrase IX
Keywords: PET; CAIX; Renal Cancer; diagnosis
MeSH Terms: conditions — Neoplasms; Kidney Neoplasms; Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Experimental: CAIX-PET/CT: Each participant receives a single intravenous injection of CAIX-PET/CT, and undergo PET/CT imaging within the specified time.

SUMMARY:
To evaluate the efficacy of targeted CAIX-specific probe PET imaging in the diagnosis and staging of kidney cancer, as well as to assess its role in prognosis prediction and treatment evaluation for kidney cancer.

DETAILED DESCRIPTION:
Images will be analyzed by at least two physicians with extensive experience in nuclear medicine and radiological diagnostics. Regions of interest (ROIs) will be delineated for the lesion tissues to measure volume and SUV values. The interpreted PET/CT imaging results will be compared to the corresponding histopathological results of the lesions (obtained through biopsy or surgery) and will be used as the reference standard. We will employ McNemar's test to compare the sensitivity, specificity, accuracy, positive predictive value, and negative predictive value of targeted CAIX PET/CT imaging and enhanced CT in primary tumors, metastatic lymph nodes, and distant metastatic lesions.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary participation with the patient or their legal representative able to sign the informed consent form.
2. Adult patients (age between 18 and 75 years), regardless of gender.
3. Patients with clinically suspected or confirmed primary kidney cancer (supporting evidence includes imaging data and histopathological examination; specific case types include clear cell carcinoma, papillary renal cell carcinoma, and chromophobe renal cell carcinoma) who agree to undergo histopathological examination (if not already performed prior to imaging).
4. Patients must have undergone enhanced CT, with the enhanced CT examination conducted within 2 weeks prior to enrollment.
5. ECOG performance status score of 0-3.
6. Laboratory parameters must meet the following criteria:

   1. ALT and AST must not exceed 3 times the upper limit of normal; BUN and creatinine must not exceed 1.5 times the upper limit of normal.
   2. Hematological parameters: 2 x 10^9/L ≤ WBC ≤ 2 x 10^10/L, PLT ≥ 80 x 10^9/L, Hb ≥ 80 g/L.
7. Willing and able to comply with follow-up visits, treatment plans, and related laboratory examinations.

Exclusion Criteria:

1. Pregnant or breastfeeding patients (all women of childbearing age must undergo pregnancy testing during the screening phase, such as a urine pregnancy test or blood HCG test, to confirm their pregnancy status).
2. Patients or their legal representatives who are unable or unwilling to sign the informed consent form.
3. Acute systemic diseases and electrolyte imbalances.
4. Patients unable to complete the PET/CT examination (including those unable to lie flat, those with claustrophobia, radiophobia, etc.).
5. Researchers believe that the patient has poor compliance or has other factors making them unsuitable for participation in this study.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. Adult patients (age between 18 and 75 years), regardless of gender.
  2. Patients with clinically suspected or confirmed primary kidney cancer (supporting evidence includes imaging data and histopathological examination; specific case types include clear cell carcinoma, papillary renal cell carcinoma, and chromophobe renal cell carcinoma) who agree to undergo histopathological examination (if not already performed prior to imaging).
  3. Patients must have undergone enhanced CT, with the enhanced CT examination conducted within 2 weeks prior to enrollment.
  4. ECOG performance status score of 0-3.
  5. Laboratory parameters must meet the following criteria:
     1. ALT and AST must not exceed 3 times the upper limit of normal; BUN and creatinine must not exceed 1.5 times the upper limit of normal.
     2. Hematological parameters: 2 x 10^9/L ≤ WBC ≤ 2 x 10^10/L, PLT ≥ 80 x 10^9/L, Hb ≥ 80 g/L.
Sampling Method: Non-Probability Sample
Enrollment: 113 (Estimated)
Dates: Start 2025-05-09 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Evaluate the clinical diagnostic efficacy | 3 Months
  To evaluate the clinical diagnostic efficacy (sensitivity, specificity, accuracy) of targeted CAIX PET/CT imaging in the diagnosis and staging of kidney cancer

SECONDARY OUTCOMES:
Assess the clinical added value | 6 Months
  To assess the clinical added value of targeted CAIX PET/CT molecular imaging technology in the diagnosis and staging of kidney cancer by comparing it with enhanced CT.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Xiamen University, Xiamen, Fujian 361000, Xiamen, China

IPD SHARING:
Plan to Share IPD: No